CLINICAL TRIAL: NCT00528138
Title: Prospective Study Comparing Hyperbilirubinemia, CRP, White Blood Cell Count, and Other Clinical Parameters for the Preoperative Diagnosis of Perforated Acute Appendicitis
Brief Title: Hyperbilirubinemia in Acute Appendicitis as a Predictor of Perforation
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Marcelo A. Beltran, Hospital De La Serena
Other Study IDs: HLS-0045-07-07
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Perforated Appendicitis
Keywords: Appendicitis; Hyperbilirubinemia; CRP; Values of bilirubin; Values of liver function test; Values of white blood cells; Values of CRP
MeSH Terms: conditions — Appendicitis; Hyperbilirubinemia | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Simple appendicitis
  Interventions: Other: Laboratory Test
- 2: Perforated appendicitis
  Interventions: Other: Laboratory Test

INTERVENTIONS:
Other: Laboratory Test — CRP, white blood cell count, hepatic function tests

SUMMARY:
It has recently been published that hyperbilirubinemia is a reliable marker for the preoperative diagnosis of perforated acute appendicitis.

The investigators believe, based on their own previous publications, that C-reactive protein (CRP) with or without a white blood cell count and some other clinical parameters, are more specific markers for the preoperative diagnosis of perforated acute appendicitis.

The purpose of this study is to prospectively compare the specificity and sensitivity of hyperbilirubinemia CRP, white blood cell count and other clinical parameters for the preoperative diagnosis of acute appendicitis.

DETAILED DESCRIPTION:
* Previously validated appendicitis score
* Time from onset of symptoms to diagnosis and to surgery
* Laboratory values: WBC, CRP, liver function test
* SIRS values
* Preoperative and postoperative diagnosis
* Length of hospital stay
* Postoperative complications
* Biopsy results

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for appendectomies for acute appendicitis at the emergency unit of our institution
* Patients older than 15 years of age to 100 years of age

Exclusion Criteria:

* Appendectomy performed incidentally or for other indications
* Patients younger than 15 years of age
* Alcoholism
* A history of viral hepatitis
* Gilbert's disease
* Dubin Johnson syndrome
* BRIC (benign recurrent intra-hepatic cholestasis) and other documented biliary
* Hemolytic or liver diseases associated with hyperbilirubinaemia

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of having acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltran, MD, Principal Investigator — Hospital de La Serena; Rodrigo Barrera, MD, Study Director — Hospital de La Serena
Locations (1):
- Hospital De La Serena - Emergency Unit, La Serena, Coquimbo Region, Chile